CLINICAL TRIAL: NCT01659684
Title: Evaluation of the Safety and Efficacy of Standard Intravenous Immunoglobulins in Pregnant Women With Primary Cytomegalovirus Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Onlus Camillo De Lellis (Other)
Collaborators: Regione Abruzzo, Italy (Unknown); Azienda Sanitaria Locale di Pescara (Other)
Responsible Party: Principal Investigator, Dr. Giustino Parruti, MD, PhD, Azienda Sanitaria Locale di Pescara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IVIG-001
Record Dates: First submitted 2012-08-01; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Cytomegalovirus Congenital Infection
Keywords: congenital CMV infection; standard immunoglobulins; immunoglobulin therapy; IgG CMV avidity index; Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- standard intravenous immunoglobulin (Experimental): Single arm evaluation of neurological consequences of congenital CMV infection in comparison with historical untreated controls.
  Interventions: Biological: standard intravenous immunoglobulin

INTERVENTIONS:
Biological: standard intravenous immunoglobulin — Human standard intravenous immunoglobulin (IVIG), 0.5 g/Kg of body weight, monthly after confirmation of primary gestational CMV infection

SUMMARY:
Because the potential benefit of standard intravenous immunoglobulins (IVIG) - obtained from unselected donor pools including a varying proportion of donors previously exposed to CMV - has not yet been explored in pregnant women, the investigators performed a longitudinal prospective study on the possible efficacy of IVIG for prevention or therapy of fetal CMV infection.

DETAILED DESCRIPTION:
Human IVIG are offered monthly to consecutive enrolled pregnant women with confirmed primary CMV infection at any stage, for the prevention and treatment of fetal CMV infection. Primary infection is defined by positive CMV IgM antibodies with absent or low titres of CMV IgG antibodies, and either low (<40%) CMV IgG avidity indexes with positive CMV IgM AND IgG antibodies. In addition women with indefinite avidity index and positive CMV DNA detection in urine and/or blood samples are also considered for treatment. Standard human intravenous immunoglobulins were chosen for their safety and efficacy, well documented in other settings. IVIGs were used to perform all of the infusions in the study, undiluted after reconstitution, in accordance with instructions of the manufacturer. We chose to perform IVIG infusions using 0.5 g/Kg of body weight, to make sure that a dose of specific CMV IgG at least comparable with that carried by HIG were infused at each time point. Infusions last 4 to 5 hours, using a double lumen line to infuse approximately 1500 mL of either 5% glucose or saline solution in parallel with the undiluted IVIG preparation, to reduce the risk of infusion reactions.

CMV IgG and IgM antibodies and IgG avidity indexes are assayed before and after each IVIG infusion, within 15 minutes. Quantitative CMV DNA is amplified from whole blood and urine samples from pregnant women and neonates, using the Real-Time PCR, and on samples of amniotic fluid from women who required amniocentesis. The newborns will be followed for five years after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with confirmed primary CMV infection at any stage of gestation.

Exclusion Criteria:

* Pregnant women with falsely positive CMV IgM antibodies or high (>40%) CMV IgG avidity indexes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Prevention of neurological damage due to Cytomegalovirus congenital infection | Neonates will be followed for 5 years, that is the estimated period of time over which late neurological manifestations may ensue
  Number of infected newborns with neurological deficits divided by the total number of infected newborns

SECONDARY OUTCOMES:
Evaluate safety of aspecific immunoglobulins in pregnant women with primary CMV infection | Participants are followed during the infusion period, an expected average of 5 hours; possible minor side-effects are searched for at each follow up visit
  Number of women with symptoms or adverse events during infusions divided by the total number of treated women

CONTACTS AND LOCATIONS:
Overall Officials: Giustino Parruti, MD, PhD, Principal Investigator — Azienda Sanitaria Locale di Pescara
Locations (1):
- Infection Disease Unit, Pescara General Hospital, Pescara, Italy, Pescara, Abruzzo, Italy